CLINICAL TRIAL: NCT02968966
Title: Pathophysiologie Basierte Therapie Von früh Beginnenden Epileptischen Enzephalopathien
Brief Title: Pathophysiology Based Therapy of Early Onset Epileptic Encephalopathies
Acronym: EE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patients recruited
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKF 357-0-0
Record Dates: First submitted 2016-11-16; First posted 2016-11-21 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Seizure, Epileptic
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Intervention Model Description: Treatment A - if no positive response: Treatment B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy regime (Experimental): Two medical drugs will be administered in a predefined order (1. Phenhydan® (Phenytoin), 2. Lacosamide (Vimpat®) to investigate whether this enables an effective reduction of seizures in early onset epileptic encephalopathies..
  Interventions: Other: Therapy regime

INTERVENTIONS:
Other: Therapy regime — Patient will receive Phenytoin, if no success is obtained, Vimpat is given. In case of success after one of the treatments, the endpoint is reached. Success is defined as reduction of seizures to 50% compared to baseline.
  Other Names: two medical products given in a predefined order

SUMMARY:
Genetic epileptic encephalopathies (EEs) are a group of very rare and severe, pharmaco-resistant epilepsy forms characterized by an early onset, e.g. first years of life, and an often severe developmental delay. Genetic defects were found in different ion channels such as potassium or sodium channels explaining well the pathological neuronal hyperexcitability leading to seizures. Further mutations were also found in proteins relevant for cell structure, DNA/RNA processing or the synaptic vesicular metabolism. Specific and individualized therapies have not been established neither in the clinical routine nor in controlled studies. The goal of this monocentric non-blinded non-placebo controlled phase IIb study is the evaluation of the effectivity of anticonvulsive drugs specifically working on the ion channels defective in some subtypes of EEs in order to establish a standard and individualized therapy for these rare diseases based on the specific genetic defect.

DETAILED DESCRIPTION:
During the study, the sodium channel blockers phenytoin and lacosamide and the potassium channel blocker kinidinsulfate will be given under standardized conditions to patients with an early onset and pharmaco-resistant genetic epilepsy with and without mutations in the potassium channels KCNT1 and KCNQ2 and the sodium channel gene SCN2A. The primary endpoint will be a significant seizure reduction under trial medication compared to baseline. Secondary endpoints will be the improvement of electroencephalographic characteristics of the respective EEs.

ELIGIBILITY:
Inclusion Criteria:

* highly active epilepsy (≥ 1 seizure per day)
* epilepsy with onset 0-3 months of age
* pharmaco-resistant epilepsy (2 or more standard anticonvulsive medications tried before)
* recently max. two stable anticonvulsive drugs for minimum 4 days before study start
* patients under continuous monitoring control
* patients younger than 1 year of age

Exclusion Criteria:

* high grade cardial rhythm disorders
* severe liver, renal and electrolyte blood parameter changes
* metabolic or lesional origin of epilepsy (metabolic screening results and cranial MRI available)
* parallel participation in other studies (must be finished two month before study start)
* missing informed consent

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Reduction of seizures | one week
  Reduction of epileptic seizures within one treatment phase to 50% compared to baseline

SECONDARY OUTCOMES:
Reduction of seizures stratified for genetic background | one week
  Reduction of epileptic seizures within one treatment phase to 50% compared to baseline stratified for three gene mutations
Reduction of epileptic activities or suppression phases | one week
  Reduction of epileptic activities or suppression phases in EEG

CONTACTS AND LOCATIONS:
Overall Officials: Markus Wolff, Dr., Principal Investigator — University Children's Hospital Tübingen
Locations (1):
- Universtiy Hospital, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Synopsis — http://www.medizin.uni-tuebingen.de/kinder/de/abteilungen/cpcs/projekte/